CLINICAL TRIAL: NCT03109418
Title: Intraoperative Low-dose Ketamine Infusion for Patients With Obstructive Sleep Apnea: A Prospective, Randomized, Controlled, Double-Blind Study
Brief Title: Intraoperative Low-dose Ketamine Infusion for Patients With Obstructive Sleep Apnea
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Peter A. Nagi, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: F160224001
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Results first posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Sleep Apnea; Obstructive Sleep Apnea; Postoperative Complications
Keywords: Ketamine; Postoperative morbidity
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Postoperative Complications | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Group (Placebo Comparator): OSA patients will receive standard inhaled anesthesia with normal saline infusion
  Interventions: Procedure: Control
- Ketamine Group (Active Comparator): OSA patients receiving standard inhaled anesthesia combined with a low-dose ketamine infusion.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — OSA patients receiving standard inhaled anesthesia combined with a low-dose ketamine infusion in which dosage will be based on ideal or adjust body weight
  Other Names: Ketalar
  Arms: Ketamine Group
Procedure: Control — OSA patients receiving standard inhaled anesthesia combined with normal saline
  Arms: Control Group

SUMMARY:
The aim of this study is to substantially reduce overall postoperative morbidity and mortality associated with obstructive sleep apnea.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) affects millions of people in the U.S., and currently, there is not a well-established, general anesthetic technique that clearly decreases the risk of postoperative respiratory complications in these patients. If OSA patients have significantly decreased postoperative opioid requirements and improved recovery profiles in the PACU, the protocol could have significant implications in defining future standardized general anesthesia recommendations for patients with this disease. Ultimately, the aim of this study is to substantially reduce overall postoperative morbidity and mortality associated with obstructive sleep apnea. The objective of this study is to compare the postoperative recovery profile of OSA patients receiving standard Sevoflurane inhaled anesthesia with normal saline infusion versus Sevoflurane combined with a low-dose ketamine infusion.

ELIGIBILITY:
Inclusion Criteria:

* aged 19-100
* scheduled to undergo general ENT or Orthopedic Surgery
* diagnosis of obstructive sleep apnea as confirmed by sleep study or deemed high risked for obstructive sleep apnea by clinical predictors (greater than 4 clinical predictors of obstructive sleep apnea as described by STOP BANG ).

Exclusion Criteria:

* positive pregnancy test
* ASA > III
* history of alcohol or narcotic abuse in last 90 days
* significant cardiovascular or respiratory disease (baseline oxygen saturation below 92%)
* significant psychiatric or neurologic disease
* history of significant hepatic or renal disease (baseline creatinine>1.5)
* history of allergy or contraindication to anesthetic agents or ketamine including patients with increased ICP
* increased IOP
* severe arrhythmias
* history of delirium
* history of hallucinations
* history of psychosis
* history of uncontrolled seizures
* potential risk for malignant hyperthermia (family history)
* history of difficult intubation that would preclude standard induction of anesthesia
* prisoners
* persons who are mentally impaired
* non-English speakers

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Nagi, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Department of Anesthesiology and Perioperative Medicine, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants were excluded prior to randomization due to the following reasons:
  1. The patient was experiencing on-going neurological issues and was therefore removed from the study prior to randomization.
  2. The patient missed his/her own surgery date.
  3. The patient ended up having outpatient surgery, and was therefore excluded.
Period: Overall Study
Arm/Group | Control Group | Ketamine Group
Started | 2 | 4
Completed | 2 | 3
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Ketamine Group | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 1 | 1
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Males | 2 | 2 | 4
  Female | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 2 | 2 | 4
  African-American | 0 | 1 | 1
  Hispanic/Latino | 0 | 0 | 0
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores
Description: Visual Analog Scale pain rating
Time Frame: up to 24 hours postoperatively
Population: Study was terminated. Data was not collected.
Arm/Group | Control Group | Ketamine Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Patient Satisfaction Score
Description: Patients will rate their quality of anesthesia services
Time Frame: At 24 hrs post-op
Population: Participants were not analyzed due to study being terminated. Data was not collected.
Arm/Group | Control Group | Ketamine Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Control Group | Ketamine Group
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 0/2 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-07-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT03109418/Prot_SAP_000.pdf